CLINICAL TRIAL: NCT03833401
Title: Dental Pulp Regeneration for Root Canals by Autologous Tissue Transplantation
Brief Title: Dental Pulp Regeneration by Autologous Tissue Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Mo K. Kang, DDS, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-000077
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Dental Pulp Regeneration

STUDY DESIGN:
Intervention Model Description: This study will involve two Arms; one serving as sham comparator, and the other arm serving as experimental (test) group.
Who Masked: Participant
Masking Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal revascularization (Sham Comparator): Root canal disinfection and revascularization without tissue transplantation. This will serve as control group.
  Interventions: Procedure: Root canal revascularization
- Autologous tissue transplantation (Experimental): Root canal disinfection will be performed and revascularization will be induced with autologous tissue transplantation.
  Interventions: Procedure: Autologous tissue transplantation

INTERVENTIONS:
Procedure: Autologous tissue transplantation — Root canal disinfection and revascularization with patient's own minced pulp tissues
  Arms: Autologous tissue transplantation
Procedure: Root canal revascularization — Root canal disinfection and revascularization without tissue transplantation
  Arms: Root canal revascularization

SUMMARY:
The purpose of this study is to develop new improved therapy for teeth that require root canals due to tooth infection or tooth inflammation. Investigators will recruit total of 50 participants from the age group 7 - 50 at the UCLA School of Dentistry Endodontic clinic. The participants will be divided into two groups, one will receive traditional therapy, which may include root canal or a procedure called "revascularization," which is a procedure trying to regrow the tissue inside the tooth. The other group of participants will receive the test treatment, which will involve harvesting of pulp tissues from the same tooth or other teeth that are planned for extraction. Investigators will prepare these tissues and place the tissues back into the cleaned root canal space with induced bleeding to allow regrowth of the tissue. For all participants, investigators will follow up after 6, 12, and 24 months in a shorter appointment, which may involve taking x-ray and clinical exam.

DETAILED DESCRIPTION:
The goal of the study is to test whether autologous pulpal mesenchymal stem cells (MSCs) is capable of de novo regeneration of pulp-dentin complex and restoration of normal pulp physiology in teeth with necrotic or inflamed pulp. This is a highly novel study that will bring the regenerative endodontic approaches to the next level. Furthermore, revascularization approaches, as delivered in today's endodontic offices, present several challenges, including lack of de novo pulp-dentin regeneration, and frequent occurrence of intracanal calcification. These findings attest to the limitation of revascularization as a regenerative endodontic procedure (REP) and necessitates advent of novel approach for functional restoration of dental pulp. The ultimate objective of the current study is to develop a new REP that allows for de novo regeneration of functional dental pulp, which can be readily performed in a chair-side manner.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants at ages of 7 - 50 y.o. presenting with a tooth diagnosed with complete or partial necrosis of the pulp or irreversible pulpitis.
* Participants presenting with donor pulp tissue, either from existing deciduous teeth or from permanent teeth treatment planned for extraction, e.g., second premolars for orthodontic extraction or third molars.
* Participants presenting with irreversible pulpitis and partial necrosis, i.e., visible pulpal tissues during access opening and canal debridement.
* Participants with immature root apices, including those with partially closed apex, that require root canal procedure.

Exclusion Criteria:

* Participants with any systemic conditions preventing routine dental procedures or requiring medication that interfere with healing or induce bleeding.
* Participants with avulsed, replanted teeth with resultant pulp necrosis.
* Participants with vertical root fracture/cracks.
* Participants with teeth that are not restorable.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in radiographic assessment for periapical inflammation | 6 months, 12 months, and 24 months
  This outcome will test the effect of treatment in either Arm on resolving periapical inflammation, which will be assessed by radiographic imaging and clinical examination. Healing of periapical inflammatory lesion will be measured by radiographic imaging to note changes in the size of pre-existing radiograph periapical lesions after the treatment.
Changes in pulpal sensibility to temperature and electric current | 6 months, 12 months, and 24 months
  This outcome will test whether the treatment in either Arm will allow revitalization of pulp tissues, by means of thermal and electrical testing of pulp vitality.
Changes in root dentin thickness of root canals | 6 months, 12 months, and 24 months
  This outcome will assess changes in root dentin thickness after treatment in either arm. We will also determine if the apical opening (foramen) will close in cases that initially present with open apices. This assessment will be based on radiographic imaging.
Changes in root length | 6 months, 12 months, and 24 months
  This outcome will assess changes in root length after treatment in either arm. This assessment will be based on radiographic imaging.
Changes of root canal calcification in teeth treated by revascularization with or without tissue transplantation | 6 months, 12 months, and 24 months
  This outcome will assess the degree of root canal calcification in teeth treated in either Arm by radiographic imaging. Degree of calcification will be measured by means of different levels of radio-opacity in routine dental X rays.

CONTACTS AND LOCATIONS:
Overall Officials: Mo Kang, DDS,PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Dentistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No